CLINICAL TRIAL: NCT05063851
Title: The Use of Memantine for Prevention of Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Carol Manning, Professor of Neurology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSR200202
Record Dates: First submitted 2021-07-23; First posted 2021-10-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Memantine hydrochloride (Experimental)
  Interventions: Drug: Memantine Hydrochloride Tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine Hydrochloride Tablets — The recommended starting dose of memantine hydrochloride/placebo is 5 mg once daily. The dose should be increased in 5 mg increments to 10 mg/day (5 mg twice daily), 15 mg/day (5 mg and 10 mg as separate doses), and 20 mg/day (10 mg twice daily). The minimum recommended interval between dose increases is one week. The dosage shown to be effective in controlled clinical trials is 20 mg/day.
  Arms: Memantine hydrochloride
Drug: Placebo — The recommended starting dose of memantine hydrochloride/placebo is 5 mg once daily. The dose should be increased in 5 mg increments to 10 mg/day (5 mg twice daily), 15 mg/day (5 mg and 10 mg as separate doses), and 20 mg/day (10 mg twice daily). The minimum recommended interval between dose increases is one week. The dosage shown to be effective in controlled clinical trials is 20 mg/day.
  Arms: Placebo

SUMMARY:
As the US population ages, the prevalence of dementia is increasing, and Alzheimer's Disease (AD) is the most prevalent one. Solving the Alzheimer's Disease (AD) epidemic is likely to require preventive therapy beginning many years before symptoms are expected to be evident in at-risk individuals. AD is caused by the dysfunction, loss of synapses, and eventual neuronal death, which may occur up to 25 years before clinical symptoms appear. This study, based off of pre-clinical data, seeks to assess whether it is feasible to use memantine hydrochloride for the prevention of Alzheimer's Disease.

DETAILED DESCRIPTION:
The use of memantine for prevention of Alzheimer's Disease (AD) is designed to assess the feasibility of the use of memantine hydrochloride for prevention of AD and provide design elements for a Phase 3 efficacy study.

Up to 128 subjects will be enrolled/screened to achieve a sample size of 32 randomized participants with a 1:1 randomization allocation. The study population will include individuals, 50-65 years of age, who are APOE4 positive with a family history of Alzheimer's Disease who meet all other eligibility criteria.

The schedule of assessments includes screening/baseline, treatment period (including titration up/down) and follow up/end of study over 101 weeks for each subject. Study efficacy assessments are the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), Montreal Cognitive Assessment (MoCA), Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL), Cognitive Function Index, Alzheimer's Disease Cooperative Study - Activities of Daily Living Prevention Instrument Activities of Daily Living - Prevention Instrument and the Clinical Dementia Rating Scale (CDR) Scale. Safety assessments include the Center for Epidemiologic Studies Depression Scale (CES-D) Vital Signs, Physical/Neurological Exam, Electrocardiogram, Blood Chemistries, Urinalysis, Medical History, Assessment of Adverse Events and Concomitant Medications, MRI and PET imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the age of 50 and 65 years at time of informed consent.
2. Have a positive family history for dementia (minimum of 1 first degree relative).
3. Previously known or documented heterozygote or homozygote ApoE ε4 allele.
4. Be able to read and write and must have adequate hearing and visual acuity to complete the psychometric tests.
5. Be otherwise healthy for their age group or medically stable with or without medication on the basis of physical examination, medical history, vital signs, and 12-lead ECG performed at screening or at baseline.
6. Have Montreal Cognitive Assessment (MOCA) score of 27 or above.
7. Have a creatinine clearance (CrCl), estimated using the Cockcroft-Gault formula, greater or equal to 30 mL/minute.

Exclusion Criteria:

1. A current clinical condition or requires a medication that raises the pH of their urine.
2. Severe renal or hepatic impairment.
3. Any other abnormality that could cause a possible cognitive deficit (including, but not limited to, vascular encephalopathy or large strokes).
4. Contraindications for MRI (e.g., prostheses, implants, claustrophobia, pacemaker) or PET imaging.
5. Neurodegenerative disorder known to cause neurocognitive decline
6. Relevant history of or current neurological disease other than preclinical AD, which may make interpretation of possible new neurological signs or symptoms difficult.
7. Clinically significant and active pulmonary, gastrointestinal, renal, hepatic, endocrine, or cardiovascular system disease
8. Ongoing cancer treatment
9. Clinically significant and active psychiatric disorder
10. Use of an investigational medical device within 3 months before the planned start of study.
11. Current participation in an interventional study with an investigational drug component.
12. Major surgery (e.g., requiring general anesthesia) within 8 weeks before screening, or will not have fully recovered from surgery, or has major surgery planned during the time the subject is expected to participate in the study.
13. Requires treatment with an AChE inhibitor or any of the following: acetazolamide, methazolamide, amantadine, ketamine, dextromethorphan.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of the use of memantine hydrochloride for prevention of Alzheimer's Disease as measured by the percentage of patients who are lost to follow-up | Baseline to 24 months
  The percentage of subjects who are lost to follow-up before completion of the protocol will be calculated, along with 95% confidence intervals. Calculations will be carried out in the entire randomized population, and by treatment arm. Loss to follow-up percentages will be compared between arms using Fisher's exact tests. Permutation tests will be used to assess if any baseline subject characteristics are associated with overall loss to follow-up percentages, or time to loss to follow-up.

SECONDARY OUTCOMES:
Summary of demographic characteristics of subjects overall, and in each arm. | Baseline to 24 months
  Permutation tests, Fisher's exact tests, or Mann-Whitney U-tests will be used depending on the data distributions observed. This is a needed design estimate for a Phase 3 efficacy trial.
Mean change in RBANS scores from baseline to end of protocol, overall and in each arm. | Baseline to 24 months
  The changes from baseline to 24 months will be calculated for each individual who completes the study. Both absolute and relative changes will be computed for each measurement. T-tests or Mann-Whitney U-test will be used to compare the change scores between arms. Additionally, since measurements are also planned at 12 months, an analysis will be performed using all available data on each subject. This analysis will use a random effects model to estimate the trajectories of change over time in each arm. The random effects model will also be used to assess the potential effect of each demographic variable on the change in RBANS. This is a needed design estimate for a Phase 3 efficacy trial.
Intraclass correlation coefficient (ICC) for longitudinal follow-up | Baseline to 24 months
  The ICC will be calculated by dividing the random effects variance in the random effects model (above) by the total variance. This is a needed design estimate for a Phase 3 efficacy trial.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Manning, PhD, Principal Investigator — Professor of Neurology; Anelyssa D'Abreu, MD, Principal Investigator — Associate Professor of Neurology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No